CLINICAL TRIAL: NCT00160628
Title: A Korean Open-label, Multi-center, Community-based Trial Assessing the Efficacy and Safety of Levetiracetam as Adjunctive Therapy in Adult Subjects With Uncontrolled Partial Epilepsy for Bridging Purpose With a Similar Study on Caucasian Epileptic Subjects
Brief Title: Open Label Safety and Efficacy Study of Levetiracetam in Korean Patients With Epilepsy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: N01099
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2010-02

CONDITIONS: Epilepsy, Partial
Keywords: Epilepsy; Partial Onset Seizures; Keppra; Levetiracetam
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam

SUMMARY:
A Korean open-label, community-based trial assessing the efficacy and safety of levetiracetam as adjunctive therapy in partial epilepsy.

Similarity with a similar study conducted in Caucasian epileptic subjects will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with epilepsy experiencing partial seizures, whether or not secondarily generalized.
* Subjects must present between 3 and 42 partial seizures over the three months prior to protocol Visit 1.
* Use of one (1), but no more than two (2) concomitant marketed AEDs at the time of trial entry.

Exclusion Criteria:

* Subjects on felbamate with less than 18 months exposure.
* Subjects on vigabatrin, whose visual field has not been assessed as per recommendation of the manufacturer, i.e. every 6 months.
* Presence of known pseudoseizures within the last year.
* Presence of progressive cerebral disease, any other progressively degenerative neurological disease, or any cerebral tumors.
* Uncountable seizures (clusters) or history of convulsive status epilepticus within the last five years.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-03; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
To evaluate efficacy of levetiracetam in community based practice (seizure frequency per week over 16 weeks).

SECONDARY OUTCOMES:
To assess safety of levetiracetam

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma

REFERENCES:
- [Result] Heo K, Lee BI, Yi SD, Huh K, Kim JM, Lee SA, Shin DJ, Song HK, Lee SK, Kim JY, Lu S, Dubois C, Tonner F. Efficacy and safety of levetiracetam as adjunctive treatment of refractory partial seizures in a multicentre open-label single-arm trial in Korean patients. Seizure. 2007 Jul;16(5):402-9. doi: 10.1016/j.seizure.2007.02.011. Epub 2007 Mar 19. PMID 17369059